CLINICAL TRIAL: NCT03645798
Title: The Effects of "Three Good Things" Positive Psychotherapy on Burnout, Turnover Intention, Job Performance, Job Satisfaction, Self-efficacy, Coping Styles, Resilience and Blood Cortisol of Chinese Nurses
Brief Title: The Effects of "Three Good Things" Positive Psychotherapy on Nurses' Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Yufang Guo, Principal Investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20150131
Record Dates: First submitted 2018-08-16; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Burnout Syndrome; Nurse's Role
Keywords: burnout; turnover intention; job performance; job satisfaction; resilience; self-efficacy; coping style; cortisol; nurse
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: A randomized, controlled trial was conducted for 73 nurses from The Second Xiangya Hospitcal of Central South University (33 in the experimental group, 40 in the control group). The experimental group received a Wechat-based six-month "three good things" positive psychotherapy from August 2015 to January 2016, while the control group only received normal psychological instruction from the hospital.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Three good things" therapy group (Experimental): The experimental group received a six-month Wechat-based"three good things" positive psychotherapy from August 2015 to January 2016. Participants were directed to record three good things that went well each day. These things could be minor, ordinary, or important. Next to each good things, participants were required to answer the question:" Why did this good thing happen"?
  Interventions: Behavioral: "Three good things" therapy
- Normal psychological instruction group (Other): The control group only received normal psychological instruction from the hospital
  Interventions: Behavioral: Normal psychological instruction

INTERVENTIONS:
Behavioral: "Three good things" therapy — To maintain an emphasis on the positive experience, participants were directed to record three good things that went well each day. These things could be minor, ordinary, or important. Next to each good thing, participants were required to answer the question: "Why did this good thing happen?"
  Arms: "Three good things" therapy group
Behavioral: Normal psychological instruction — Normal psychological instruction is a convenient method set by the hospital. Nurses who have stress or psychological problem could find help through this intervention. It was delivered by psychologists.
  Arms: Normal psychological instruction group

SUMMARY:
A randomized, controlled trial was conducted for 73 Chineses nurses from The Second Xiangya Hospitcal of Central South University (33 in the experimental group, 40 in the control group). The experimental group received a six-month Wechat-based "three good things" positive psychotherapy from August 2015 to January 2016, while the control group only received normal psychological instruction from the hospital. A socio-demographic sheet, Malsach Burnout Inventory-General Survey, the Turnover Intention Scale, The Job Satisfaction Scale, The Job Performance Scale, General Self-efficacy Scale, The Trait Coping Style Scale (TCSS), The Connor-Davidson Resilience Scale (CD-RISC) were used to collect data prior to and immdediately after the intervention. The blood cortisol was also evaluated prior to and immdediately after the intervention. SPSS 23.0 was used for data analysis. Descriptive statistics, ANOVA, Chi-square test, repeated-measures analysis and T-test were employed to analyse the effect of "three good things" intervention on nurse burnout. We hypothesis that the "three good things" positive psychotherapy could alleviate nurses' burnout, turnover intention, improve their job performance, job satisfaction, self-efficacy, resilience, introduce nurses' to use positive coping strategies to overcome adversities. Moreover, their blood cortisol would be reduced after the intervention.

DETAILED DESCRIPTION:
Study design and sample In the present study, we used a randomized, controlled design to assess the effect of "three good things" positive psychotherapy from August 2015 to January 2016. Measures were administered before (T0) and immediately after (T1) the intervention.

The study sample were nurses recruited from one three-level general hospital in Changsha, Hunan, China. The sample size calculation was conducted via PASS statistical software (NCSS LCC, East Kaysville, UT, USA) . The effect size was 0.67, power was 0.80, and margin of error type Ⅰ was 0.05. Accordingly, the sample size was 64. Stochastic tables' law was used for group division. A total of 193 nurses completed the MBI-GS, and 102 nurses who met the inclusion criteria were randomly selected for the study. However, only 73 completed the study, with 33 in the experimental group and 40 in the control group.

Instruments A socio-demographic questionnaire, the Maslach Burnout Inventory-General Survey (MBI-GS), the turnover intention questionnaire, the Job Performance scale, the Job Satisfaction scale, the General self-efficacy Scale, the CD-RISC and the Trait Coping Style Scale were used to collect the data. The blood cortisol was also collected. The detail instruction of these scales could be found at Outcome Measures section.

Ethical consideration This study was approval by The Institutional Review Board (IRB) of Xiangya Nursing School, Central South University. Participants were informed about the objectives and procedures of the study before they began the survey. All data were held confidential. Only the research team could access the data.

Data analysis Data analysis was performed using SPSS 22.0 (SPSS Inc., Chicago, IL, USA). Descriptive statistics was used to describe demographic data, burnout, turnover intention, job performance, job satisfaction, self-efficacy, resilience, coping style and cortisol. Generalized repeated-measures analysis of variance (ANOVA) was used to demonstrate the effect of intervention and time-intervention interaction.

ELIGIBILITY:
Inclusion Criteria:

* registered nurses or licenced practical nurses
* who provided direct care to residents
* who's MBI-GS score were no less than 1.5
* who didn't take any hormone therapy
* were Chinese speakers.

Exclusion Criteria:

* student nurses
* who suffered from diseases that influence their hormone levels
* who participated similar studies
* who had no interest in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
The Maslach Burnout Inventory-General survey (MBI-GS) was used to assess the change of burnout from baseline to six months later. | The MBI-GS was used to assess nurses' burnout prior to and immediately after the intervention.
  This scale was developed by Maslach and Jackson (1981) and consists of 16 items over three metrics: emotional exhaustion (EE, five items), cynicism (CY, five items) and reduced professional efficacy (RPE, six items). The items were scored on a Likert scale from 0 (never) to 6 (everyday) (Schaufeli et al. 1996). The higher the scores on the three metrics, the higher level of burnout indicated. The Chinese version of the MBI-GS, developed by Li & Shi (2003), also has a good validity and reliability. In this study, Cronbach alpha coefficients for EE, CY and RPE were 0.93, 0.83 and 0.82, respectively.

SECONDARY OUTCOMES:
The Connor-Davidson Resilience Scale (CD-RISC) | The CD-RISC was used to assess nurses' resilience prior to and immediately after the intervention.
  The CD-RISC was used to measure nurses' resilience level (Connor & Davidson 2003). This scale comprises 25 items over three metrics (tenacity, strength and optimism) that assess resilience or capacity to change and cope with adversity. Nurses were asked to rate each item with reference to the previous month. A 5-point Likert scale was used (0 = not true at all, 4 = true all the time.). The total score ranges from 0 to 100, with higher scores indicating higher levels of resilience. The Cronbach alpha coefficients of the Chinese version were 0.91 for the total score, 0.88, 0.80 and 0.60 for the three factors (Yu & Zhang 2007).
The General Self-efficacy Scale | The General Self-efficacy Scale was used to assess nurses' self-efficacy prior to and immediately after the intervention.
  Self-efficacy was defined as the average score on the General Self-efficacy Scale. The scale is a single-dimension scale with 10 questiona. Each question is assigned points from 1 to 4, and the final score is the total score of the 10 questions. The Chinese versison also has a good validity and reliability with a Cronbach alpha is 0.88.
The Trait Coping Style Scale (TCSS) | The TCSS was used to assess nurses' coping styles prior to and immediately after the intervention.
  The TCSS consists of 20 items over two metrics: positive coping style (PCS, 10 items) and negative coping style (NCS, 10 items). The items were scored on a five-point Likert scale from 1 to 5. The final scores of PCS and NCS were the total scores of their items. The Cronhach alpha coefficients of the two metrics were 0.70 and 0.69, respectively.

OTHER OUTCOMES:
The Turnover Intention Scale | The Turnover Intention Scale was used to assess nurses' turnover intention prior to and immediately after the intervention.
  The Turnover Intention Scale was developed by Michaels and Spector (1982). The Chinese version was translated by Li and Li (2000). It includes three metrics ( the possibility to resign the job, the possibility to find another job and the possibility to get another job) and 6 items. A 4-Likert scale from 1 (never) to 4 (always) was used to score each item. The higher the score was, the stronger the turnover intention is.
The Job Satisfaction Scale | The Job Satisfaction Scale was used to assess nurses' job satisfaction prior to and immediately after the intervention.
  The Job Satisfaction Scale, developed by Tao et al. (2009), includes 38 items. A 5-Likert scale from 1 (totally agree) to 5 (totally disagree) were used to score each item. The total score of job satisfaction ranges from 38 to 190, with higher score indicating higher levels of job satisfaction. The Cronbach alpha was 0.783 in this study.
The Job Performance Scale | The Job Performance Scale was used to assess nurses' job performance prior to and immediately after the intervention.
  The Job Performance Scale consists 16 items and 3 metrics (job denotion, task performance and interpersonal promotion). A 6-Likert scale from 1 to 6 was used to score nurses' job performance. The final score of the three metrics were the total score of their items. The Cronbach alpha of the three metrics in this study were 0.842, 0.904 and 0.927, respectively.
The blood cortisol | The blood was used to assess nurses' cortisol level prior to and immediately after the intervention.
  The blood sample were collected on a day during the third to the tenth day of the menstrual cycle. Participants were instructed not to eat or drink anything other than water, and not to undertake any strenuous exercise 2 h or smoking 30 min before a blood sample was taken. Five trained researchers drew the blood samples between 7am-9am at an experimental lab. Nurses were instructed to take a blood sample at their convenient time. Blood was collected using vacuum blood collection tubes (Hubei Jin Xing Technology Co. Wuhan) and sent to an endocrinology laboratory for biochemical analysis at no cost to the participants (Endocrinology Laboratory, The Second Xiangya Hospital of Central South University, Dr. Z.X. Gui). Blood samples were centrifuged at 4000 rpm for 2 min in order to get a clear supernatant. Blood cortisol was measured using an immunoassay with chemiluminescence detection (ADVIA Centaur XP Immunoassay System, Siemens, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Jingping Zhang, Study Director — Cental South University
Locations (1):
- Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
The nurses were agreed to participate in this study. However, they personal informations, such as name, age and identification number, were collected in this study, they didn't want others to access the data.

REFERENCES:
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Cameron F, Brownie S. Enhancing resilience in registered aged care nurses. Australas J Ageing. 2010 Jun;29(2):66-71. doi: 10.1111/j.1741-6612.2009.00416.x. PMID 20553536
- [Background] Bobbio A, Manganelli AM. Antecedents of hospital nurses' intention to leave the organization: A cross sectional survey. Int J Nurs Stud. 2015 Jul;52(7):1180-92. doi: 10.1016/j.ijnurstu.2015.03.009. Epub 2015 Mar 18. PMID 25863657
- [Background] Duffield CM, Roche MA, Homer C, Buchan J, Dimitrelis S. A comparative review of nurse turnover rates and costs across countries. J Adv Nurs. 2014 Dec;70(12):2703-12. doi: 10.1111/jan.12483. Epub 2014 Jul 23. PMID 25052582
- [Background] Goh YS, Lopez V. Job satisfaction, work environment and intention to leave among migrant nurses working in a publicly funded tertiary hospital. J Nurs Manag. 2016 Oct;24(7):893-901. doi: 10.1111/jonm.12395. Epub 2016 May 12. PMID 27169747
- [Background] Gringart E, Jones B, Helmes E, Jansz J, Monterosso L, Edwards M. Negative stereotyping of older nurses despite contact and mere exposure: the case of nursing recruiters in Western australia. J Aging Soc Policy. 2012;24(4):400-16. doi: 10.1080/08959420.2012.735170. PMID 23216348
- [Background] Harker R, Pidgeon AM, Klaassen F, King S. Exploring resilience and mindfulness as preventative factors for psychological distress burnout and secondary traumatic stress among human service professionals. Work. 2016 Jun 8;54(3):631-7. doi: 10.3233/WOR-162311. PMID 27286075
- [Background] Havaei F, MacPhee M, Dahinten VS. RNs and LPNs: emotional exhaustion and intention to leave. J Nurs Manag. 2016 Apr;24(3):393-9. doi: 10.1111/jonm.12334. Epub 2015 Sep 8. PMID 26347211
- [Background] Hudgins TA. Resilience, job satisfaction and anticipated turnover in nurse leaders. J Nurs Manag. 2016 Jan;24(1):E62-9. doi: 10.1111/jonm.12289. Epub 2015 Mar 17. PMID 25782613
- [Background] Jordan K, Fenwick J, Slavin V, Sidebotham M, Gamble J. Level of burnout in a small population of Australian midwives. Women Birth. 2013 Jun;26(2):125-32. doi: 10.1016/j.wombi.2013.01.002. Epub 2013 Feb 8. PMID 23395361
- [Background] Lagerlund M, Sharp L, Lindqvist R, Runesdotter S, Tishelman C. Intention to leave the workplace among nurses working with cancer patients in acute care hospitals in Sweden. Eur J Oncol Nurs. 2015 Dec;19(6):629-37. doi: 10.1016/j.ejon.2015.03.011. Epub 2015 Apr 29. PMID 25935682
- [Background] Mcmillan K, Butow P, Turner J, Yates P, White K, Lambert S, Stephens M, Lawsin C. Burnout and the provision of psychosocial care amongst Australian cancer nurses. Eur J Oncol Nurs. 2016 Jun;22:37-45. doi: 10.1016/j.ejon.2016.02.007. Epub 2016 Mar 22. PMID 27179891
- [Background] Perry L, Gallagher R, Duffield C, Sibbritt D, Bichel-Findlay J, Nicholls R. Does nurses' health affect their intention to remain in their current position? J Nurs Manag. 2016 Nov;24(8):1088-1097. doi: 10.1111/jonm.12412. Epub 2016 Jul 14. PMID 27411513

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT03645798/Prot_SAP_000.pdf